CLINICAL TRIAL: NCT04549220
Title: Seroepidemiology of Maternally-derived Antibody Against Group B Streptococcus (GBS) in Mulago/Kawempe Hospitals Uganda
Brief Title: Serosurveillance Study of Maternally Derived Anti-GBS Antibody
Acronym: ProGreSs
Status: Active, not recruiting | Type: Observational
Sponsor: St George's, University of London (Other)
Collaborators: MU-JHU CARE (Other); MRC/UVRI and LSHTM Uganda Research Unit (Other)
Responsible Party: Sponsor
Other Study IDs: 17.0018
Record Dates: First submitted 2020-09-08; First posted 2020-09-16 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Group B Streptococcus Carrier in Childbirth; Group B Streptococcal Infection, Late-Onset; Group B Streptococcal Infection, Early-Onset; Group B Streptococcus Neonatal Sepsis; Group B Strep Infection
MeSH Terms: conditions — Streptococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Delivery (Birth) Cohort: All women greater than or equal (≥) to 18 years of age and emancipated minors aged between 14 and 17 years of age delivering a live infant or stillbirth at Kawempe Referral Hospital over a 6-month pilot phase will be invited to participate in the study until a sample size of at least 5000-6000 women is achieved.
- Active Surveillance Cohort: This is expected to improve capacity for managing and investigating infants <3 months of age presenting with suspected sepsis at Kawempe Neonatal Intensive Care Unit (NICU), Postnatal Ward, and Acute Paediatric Wards and Mulago Hospital Paediatric Acute Care Unit, through provision of supplies for blood culture, CSF culture and nasopharyngeal swabs. Mothers/caretakers of Neonates that are diagnosed with GBS through this active case surveillance will be invited to participate in the study and will be enrolled following written informed consent.

SUMMARY:
Globally, neonatal mortality remains unacceptably high, with little change in the death rate in the first 28 days of life since 1990, despite reductions in under-5 mortality of up to 50% over the same period. In 2014, neonatal deaths accounted for 44% of all deaths in children under 5 with neonatal infection accounting for over a third of all deaths. Group B Streptococcus (GBS) is a major cause of septicemia and meningitis in infants globally and a cause of severe adverse neurodevelopmental outcomes in up to 50% of meningitis survivors. It can also lead to sepsis in pregnant women. GBS acquisition occurs through vertical transmission in 15%-50% of infants born to a vaginally/rectally colonized mother. Maternal colonization is a prerequisite for early onset (EO) and a risk factor for late onset (LO) disease.

Our proposal will provide these critical data in Uganda (a country with high neonatal disease burden) in a 12 month pilot study to determine: the burden of GBS disease in a cohort of mother/infant pairs and establish an active surveillance platform for monitoring of early and late onset neonatal infection in term and preterm infants in Uganda and compare this to the burden known for other African countries. This provides essential data on GBS disease outcomes from a high-HIV burden African cohort reflecting the usual standard of care in a low income, highly deprived urban environment. This pilot study will establish minimum disease estimates in the Ugandan cohort to determine the feasibility of a cohort study over three years to determine the level of antibody against GBS in cord blood from pregnancies where women are GBS colonized and non-colonized but whose infants do not develop GBS disease in the first three months of life and compare this to the level in the blood of infants who develop GBS disease. We will compare these results with those from other African countries such as South Africa to enable a robust estimate of potential sero-correlates of protection from natural infection against the most common GBS-disease-causing serotypes.

ELIGIBILITY:
Delivery (Birth) Cohort

Inclusion Criteria:

* consecutive mothers greater than or equal (≥) the age of 18 years delivering at Kawempe Hospital (live or stillbirth) and emancipated minors aged between 14-17 years of age,
* willing to stay in the area for the first three months of life or willing to travel to clinic until their child is 2 years old if their infant has known or presumed GBS infection).

Exclusion Criteria:

* Unable to give written informed consent

Active Surveillance Cohort Matching & Adjustment Criteria: (these will be applied at the analysis stage): (i) exposure to intrapartum antibiotic prophylaxis: defined as intravenous penicillin, ampicillin, cefazolin, clindamycin or vancomycin, for ≤2 hours before delivery. (ii) blood transfusion in the 30 days before delivery (iii) HIV status (iv) Maternal age (v) Infant gestational age

Min Age: 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on pregnancy
Study Population: The study will enrol pregnant women from the general population who deliver at Kawempe Hospital and follow their infants to 90 days of age.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2019-04-24 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Maternal anti-GBS antibody concentration in infants with GBS disease compared to healthy controls. | 31 October 2020
  To establish maternal anti-GBS antibody concentration in infants with GBS disease compared to healthy controls.

SECONDARY OUTCOMES:
Health-centre level active surveillance | 31 October 2020
  To establish health-centre level active surveillance for neonatal sepsis and meningitis and GBS-related stillbirths.
Neurodevelopmental outcomes | 31 October 2020
  To establish the neurodevelopmental outcomes of infants with GBS disease in Uganda up to 2 years of age.
GBS colonisation | 31 October 2020
  To determine the GBS colonisation rate and serotypes in Ugandan women at delivery

CONTACTS AND LOCATIONS:
Overall Officials: Kirsty Le Doare, Dr., Principal Investigator — St George's, University of London
Locations (1):
- MUJHU Care Ltd, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No